CLINICAL TRIAL: NCT01227837
Title: Effect of Omega 3 Supplementation on Brain Natriuretic Peptide (BNP) Serum Levels Functional Capacity and Systolic and Diastolic Function of Heart Failure Patients
Brief Title: Effect of omega3 on Congestive Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Dr Javad Kojuri, Shiraz University of medical sciences
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1388-2365
Record Dates: First submitted 2010-09-13; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-09

CONDITIONS: Heart Failure Congestive
Keywords: omega 3; CRT_AICD; congestive heart failure; CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Sham Comparator): use of placebo in control group
  Interventions: Dietary Supplement: placebo
- omega 3 (Experimental): use of omega 3 2 gr/day for 6 months
  Interventions: Dietary Supplement: omga3

INTERVENTIONS:
Dietary Supplement: placebo — placebo given to patients
  Arms: placebo
Dietary Supplement: omga3 — use of omega 3
  Arms: omega 3

SUMMARY:
In this double blinded study patients with resynchronization pacemaker- AICD were assigned to Omega3 and placebo randomly, results indicated that Omega3 had no more effect than placebo in mortality, BNP level and 6 minutes walk test.

DETAILED DESCRIPTION:
Introduction: Widely used as lipid lowering agents, Omega 3 fatty acids have been demonstrated to possess the potential to reduce the risk of cardiovascular events in patients suffering from chronic heart conditions. In this double -blinded randomized placebo-controlled clinical trial, we aim to investigate the possible beneficial effects of Omega-3 supplements on echocardiographic parameters and brain natriuretic peptide (BNP) plasma levels in patients suffering from congestive heart failure (CHF).

Methods and Materials: 100 patients with class II and III CHF, who had tri-chamber pacemaker and automated defibrillator( CRT-AICD) were initially recruited among which 70 subjects consented to participate. Subjects were randomly assigned and matched to two treatment groups. 42 patients were allocated to a two gram/day dosing of omega-3 capsule while 28 subjects were allocated to the placebo group. Demographic features and BNP plasma levels, 6-minute walk test and echocardiographic parameters of patients were recorded at baseline and at 6 months after implementation of treatment protocols. Data were further gathered and analyzed to evaluate the beneficial effects of omega-3 supplements compared to placebo.

Conclusion: Beneficial effects of Omega-3 supplementation on CHF patients were not as dramatic as initially presumed

ELIGIBILITY:
Inclusion Criteria:

* EF< 40%
* sinus rhythm
* accept randomization

  * having tri-chamber pacemaker

Exclusion criteria:

* survival less than 6 months
* class IV heart failure
* using drugs other than study protocol

Ages: 3 Months to 73 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-03

PRIMARY OUTCOMES:
BNP level | 6 months
  level of BNP in serum of patient prior and 6 months post recruitment
six minutes walk test | 6 months
  ability to walk in six minutes after and before to syudy
echocardiographic data | 6 months
  Ejection fraction Tei index Sm,Em, Am indexes of tissue doppler study

SECONDARY OUTCOMES:
mortality | 6 months
  any cardiac mortality in 6 months
hospital admission | 6 months
  any hospital admission due to cardiac problem in 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kojuri J, Ostovan MA, Rezaian GR, Archin Dialameh P, Zamiri N, Sharifkazemi MB, Jannati M. Effect of omega-3 on brain natriuretic peptide and echocardiographic findings in heart failure: Double-blind placebo-controlled randomized trial. J Cardiovasc Dis Res. 2013 Mar;4(1):20-4. doi: 10.1016/j.jcdr.2013.02.013. Epub 2013 Feb 27. PMID 24023466